CLINICAL TRIAL: NCT01615666
Title: A Composite MR Neuroimaging Marker for Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: This was never a clinical trial and should never have been approved.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2R01AG020279-06A2 (NIH); 2R01AG020279-06A2 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Frontotemporal Dementia
Keywords: Alzheimer's disease; Mild Cognitive Impairment; Frontotemporal dementia; fMRI; functional neuroimaging; Memory
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal (cheek) swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy volunteers: Healthy volunteers who will undergo functional MRI (fMRI) to obtain fMRI index
- Alzheimer's disease: Individuals with Alzheimer's disease who will undergo functional MRI (fMRI) to obtain fMRI index
- Non-Alzheimer's dementia: Individuals with Non-Alzheimer's dementia who will undergo functional MRI (fMRI) to obtain fMRI index
- Amnestic mild cognitive impairment: Individuals with Amnestic mild cognitive impairment who will undergo functional MRI (fMRI) to obtain fMRI index
- Nonamnestic mild cognitive impairment: Individuals with Nonamnestic mild cognitive impairment who will undergo functional MRI (fMRI) to obtain fMRI index

SUMMARY:
The purpose of this study is to use a functional MRI (fMRI) index to compare the brain activity of healthy volunteers to that of people with mild cognitive impairment (MCI) and Alzheimer's disease. The ultimate goal is to develop an early diagnostic tool for Alzheimer's disease.

The study hypotheses are:

1. The fMRI index will differentiate between Alzheimer's disease, non-Alzheimer's dementia, and healthy volunteers;
2. The fMRI index will distinguish participants with MCI who convert to Alzheimer's disease from those who convert to a non-Alzheimer's dementia and those who remain stable;
3. MCI participants with a lower fMRI index at baseline who convert will progress to Alzheimer's sooner than those with a higher fMRI index, and MCI participants with a faster rate of fMRI index decline who convert will have an earlier onset of Alzheimer's disease.

DETAILED DESCRIPTION:
The onset of Alzheimer's disease is insidious and the boundary between normal aging and Alzheimer's disease is blurred. In order to prevent and treat Alzheimer's disease, the investigators must be able to mark its preclinical stage, before brain damage becomes irreversible. There is a substantial body of research dealing with predictive markers of Alzheimer's disease in individuals with mild cognitive impairment (MCI). Despite these advances, however, researchers have not had enough evidence to recommend specific techniques that mark preclinical Alzheimer's disease. This new functional MRI (fMRI) index may fill this gap.

Participants will have two visits, one for memory testing and neurological examination, and one for an MRI scan. Each visit will take approximately 1½ hours. For volunteers who wish to do so, all study procedures may be completed in a single visit. Participants with MCI will be followed annually.

The investigators are currently enrolling healthy volunteers, as well as individuals with MCI (memory loss that does not significantly affect normal daily activities), Alzheimer's disease, and frontotemporal dementia (includes primary progressive aphasia).

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older (50 years of age or older for frontotemporal dementia patients)
* Normal memory, mild cognitive impairment (memory loss that does not significantly affect normal daily activities), or clinical diagnosis of Alzheimer's disease or frontotemporal dementia (includes primary progressive aphasia)
* Right-handed
* General good physical health

Exclusion Criteria:

* History of stroke or neurological disease (other than Alzheimer's disease or frontotemporal dementia)
* Seizures or head injury with loss of consciousness within the last five years
* Ferrous (magnetic) or electronic implants (due to the magnet in the MRI scanner)
* Claustrophobia

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Alzheimer's, non-Alzheimer's dementia, and mild cognitive impairment (MCI) participants recruited from the Medical College of Wisconsin/Froedtert Hospital Memory Disorders Clinic
  * MCI and healthy volunteers recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity of the MRN Index as an AD biomarker. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Jiang Li, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin, United States